CLINICAL TRIAL: NCT05541900
Title: A Conditioning Paradigm to Increase Affinity for Sacredness of Life and Decrease Experiences of Suicide-related Thoughts and Behaviors
Brief Title: A Conditioning Paradigm to Increase Affinity for Sacredness of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Military Suicide Research Consortium (Other)
Responsible Party: Principal Investigator, Anna Gai, Doctoral Candidate, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002785
Record Dates: First submitted 2022-08-29; First posted 2022-09-15 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Suicidal Ideation; Suicide, Attempted; Suicide and Self-harm; Non-suicidal Self-injury
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Suicide; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEC-Sacredness (Active Comparator): Active condition of the intervention. For the active intervention group, the three match types are as follows: (1) a self-related word paired with a life-related stimulus; (2) a sacredness of life-related stimulus paired with a pleasant stimulus; and (3) a neutral stimulus paired with a neutral stimulus.
  Interventions: Behavioral: TEC-Sacredness
- TEC-Control (Placebo Comparator): Control condition of the intervention. The control paradigm maintains the same parameters, however, all three match pairings will be neutral.
  Interventions: Behavioral: TEC-Control

INTERVENTIONS:
Behavioral: TEC-Sacredness — The participant is asked to identify and select the correct match on each trial as quickly as possible. Match pairs (i.e., a self-related word paired with a life-related stimulus, a sacredness of life-related stimulus paired with a pleasant stimulus, and a neutral stimulus paired with a neutral stimulus) are first presented to the participant. A grid is then shown containing one of the match pairs along with distraction stimuli.
  Arms: TEC-Sacredness
Behavioral: TEC-Control — The participant is asked to identify and select the correct match on each trial as quickly as possible. Match pairs (i.e., a neutral stimulus paired with a neutral stimulus) are first presented to the participant. A grid is then shown containing one of the match pairs along with distraction stimuli.
  Arms: TEC-Control

SUMMARY:
Suicide-related experiences affect millions of people every year in the United States. Through decades of research, interventions targeting these experiences have developed with varied empirical support. Many of these treatments require regular attendance to in-person sessions with a trained behavioral health professional. Limitations of in-person services have led to the development of digital-based interventions, such as Therapeutic Evaluative Conditioning (TEC). TEC is based in evaluative conditioning principles and is a brief (1-2 minutes) digital intervention designed to increase aversion to self-injurious behaviors while decreasing aversion to the self through a match game-like task. Initial assessment of the intervention demonstrated promising results although treatment effects did not remain over time. Separately, sanctification, or the process through which aspects of life are perceived as having divine character and significance, can come from a theistic or nontheistic background and does not require a belief in a God or higher power to be experienced. When something is discovered as sacred, that sacredness becomes a priority for the individual, initiating motivation to conserve what is viewed as sacred. The primary aim of the current study is to develop and test the effectiveness of an adapted version of TEC designed to increase affinity for sacredness of life and increase the connection to life as mechanisms for decreasing suicide-related experiences. Results will provide insight into the perception of sacredness of life as a potential treatment target and are foundational work in a novel approach to address the public health priority of prevention and treatment of suicide-related experiences.

DETAILED DESCRIPTION:
The present study uses an adapted version of the Therapeutic Evaluative Conditioning paradigm and principles of classical conditioning. Therapeutic Evaluative Conditioning (TEC) was designed as a brief, game-like intervention. The conditioning paradigm will follow the same structure as the original TEC intervention with specific themes modified to the current study aims. The intervention will be administered via a cloud software platform designed specifically for the administration of behavioral paradigms. Following instructions, the participant is shown three pairs of stimuli (i.e., three "matches"). In subsequent trials, one of the three matches is presented, along with non-target matches. The participant is asked to identify and select the correct match on each trial as quickly as possible. On average, each match will be presented on one-third of trials. For the active intervention group, the three match types are as follows: (1) a self-related word paired with a life-related stimulus; (2) a sacredness of life related stimulus paired with a pleasant stimulus; and (3) a neutral stimulus paired with a neutral stimulus. The control paradigm maintains the same parameters, however, all three match pairings will be neutral. Each trial presents only one possible match.

A total of 60 trials are completed in one iteration and it takes approximately 1 - 2 minutes to complete. A total of 5 iterations will be completed each week. Distraction stimuli follow the themes of the target stimuli (i.e., sacredness of life, positive stimuli, self-related words, life-related stimuli, and neutral stimuli) to add difficulty and increase the effects of the conditioning principles. For example, if the pre-determined matched pair for a trial was sacredness of life stimulus with a positive stimulus, the distraction stimuli would be either sacredness of life-related stimuli, positive stimuli, or neutral stimuli.

Pleasant and neutral stimuli will be images obtained from the International Affective Pictures System (IAPS). The sacredness of life stimuli will be generated using images from stock photo websites with free use without attribution licenses (Creative Commons Zero licenses) and words related to sacredness of life. These images and words will include both theistic and nontheistic representation of sacredness of life.

Procedures Involved:

A sample of 200 US adults (100 per group) will be recruited for the present study. All study procedures will be completed online in a location and using a device of the participant's choosing. Participants will be recruited from (1) online web forums focused on topics of self-injury or psychopathology (i.e. Reddit: r/Depression, r/SuicideWatch, r/MentalHealth; Facebook: "Suicide is real I don't want to die [help/talk], Depression/suicide, Suicide, Self Harm, I am not okay **memes&support**, Depression, Anxiety, Self Harm, Suicide Support, Depression, anxiety, and suicide, Suicide Awareness and Prevention, Support Group for Suicide, Depression, and Self Harm, Suicide Awareness, Grieving, Depression, PTSD, PP Depression, Suicide Ideation you must go), (2) email listservs for groups related to self-injury or psychopathology (i.e. listserv of the American Association of Suicidology, listserv of the Society of Clinical Psychology, Division 12 of APA, listserv of the Association of Behavioral and Cognitive Therapies, Zerosuicide listserv), and (3) from general posts on social media platforms (i.e. Facebook, Twitter, and Instagram). Postings will include a link to the screening survey. Should inclusionary criteria be met, the participant will be directed to the consent form and then to start the baseline questionnaire. Following consent, the participant will be required to provide an email address where all study contact will be made (i.e. compensation, weekly reminders, month follow-up reminder, and suicide risk outreach as needed). Participants will be provided with a unique ID number at the time of their first weekly task that they will input at the onset of each iteration of the study in order to link responses across weeks.

The experiment will be conducted fully online and will consist of assessments at baseline, weekly intervals during the treatment period, and at a month following the completion of treatment (baseline, week 1, week 2, week 3, week 4, and posttreatment). Following the completion of the baseline assessments, participants will be randomized to either the active intervention or control.

Emails will be sent on a weekly basis with links to complete each iteration of the intervention and the related questionnaires (for weeks 2 and 4 and posttreatment). Participants will receive daily email reminders for 5 consecutive days or until survey completion for that week, whichever comes first. At the end of each survey completion, participants will be given a series of mental health and suicide resources, regardless of their answers to the questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* English-language Proficiency
* History of suicide-related thoughts and behaviors and/or elevated on depressive disorder symptoms within the past month, as assessed by an elevated scored (5 or higher) and/or endorsement on Item 9 (on suicide risk) of the Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001).

Exclusion Criteria:

* Under 18
* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

PRIMARY OUTCOMES:
Perceived Sacredness of Life | After treatment completion (week 4)
  Scores on the Perceiving Sacredness of Life scale will be utilized as the main outcome for treatment targets. The Perceiving Sacredness in Life Scale assesses the extent to which an individual perceives life as sacred. The initial section of the scale lists six statements about God: theistic, deistic, pantheistic or panentheistic, agnostic, atheistic, and none of the above. This initial section is designed to orient the individual to answer the remaining 28-items (14 theistic and 14 non-theistic) based on their individual definition of God. Items are rated based on frequency of each experience and scaled from 1 - Never to 5 - Very Often. Items cover nine categories of perceiving sacredness of life, including, in general, nature and creation, time, everyday life, the journey of life, people in general, relationships with people, the self, and qualities or aspects of life. Higher scores indicate a higher perception of sacredness of life.
Perceived Sacredness of Life | One-month following treatment completion
  Scores on the Perceiving Sacredness of Life scale will be utilized as the main outcome for treatment targets. The Perceiving Sacredness in Life Scale assesses the extent to which an individual perceives life as sacred. The initial section of the scale lists six statements about God: theistic, deistic, pantheistic or panentheistic, agnostic, atheistic, and none of the above. This initial section is designed to orient the individual to answer the remaining 28-items (14 theistic and 14 nontheistic) based on their individual definition of God. Items are rated based on frequency of each experience and scaled from 1 - Never to 5 - Very Often. Items cover nine categories of perceiving sacredness of life, including, in general, nature and creation, time, everyday life, the journey of life, people in general, relationships with people, the self, and qualities or aspects of life. Higher scores indicate a higher perception of sacredness of life.
Suicide-Related Thoughts and Behaviors | After treatment completion (week 4)
  Responses on an online-version of the Self-injurious Thoughts and Behaviors Interview - Short Form will assess circumstances around previous suicidal ideation, attempts, and non-suicidal self-injury (NSSI). The SITBI-SF is a 72-item measure assessing the circumstances around previous suicidal ideation, attempts, and non-suicidal self-injury (NSSI). The SITBI-SF includes both yes/no questions on presence of suicide-related experiences as well as individual items assessing severity and other circumstances around suicide-related experiences, with higher ratings indicating more severity.
Suicide-Related Thoughts and Behaviors | One-month following treatment completion
  Responses on an online-version of the Self-injurious Thoughts and Behaviors Interview - Short Form will assess circumstances around previous suicidal ideation, attempts, and non-suicidal self-injury (NSSI). The SITBI-SF is a 72-item measure assessing the circumstances around previous suicidal ideation, attempts, and non-suicidal self-injury (NSSI). The SITBI-SF includes both yes/no questions on presence of suicide-related experiences as well as individual items assessing severity and other circumstances around suicide-related experiences, with higher ratings indicating more severity.
Modified Affect Misattribution Procedure: Implicit affinity to sacredness of life. | After treatment completion (week 4)
  A modified version of the Affect Misattribution Procedure (AMP) will be used to assess for changes in implicit attitudes on the sacredness of life. During each trial, one of the stimuli utilized in the active conditioning paradigm is presented on the screen as an emotional prime (75ms), followed by a blank screen (125ms), an ambiguous Chinese symbol (100ms) and a final blank screen. The participant is instructed to indicate whether they felt the Chinese symbol presented was "pleasant" or "unpleasant". An AMP score is calculated as the proportion of pleasant ratings within a given stimulus category rated as pleasant. For the current study, 48 trials of the AMP will be administered.
Modified Affect Misattribution Procedure: Implicit affinity to sacredness of life. | One-month following treatment completion
  A modified version of the Affect Misattribution Procedure (AMP) will be used to assess for changes in implicit attitudes on the sacredness of life. During each trial, one of the stimuli utilized in the active conditioning paradigm is presented on the screen as an emotional prime (75ms), followed by a blank screen (125ms), an ambiguous Chinese symbol (100ms) and a final blank screen. The participant is instructed to indicate whether they felt the Chinese symbol presented was "pleasant" or "unpleasant". An AMP score is calculated as the proportion of pleasant ratings within a given stimulus category rated as pleasant. For the current study, 48 trials of the AMP will be administered.
"Death/Life" Implicit Association Test. | After treatment completion (week 4)
  The d-IAT uses reaction time to measure automatic implicit associations with death and life stimuli. Procedures follow those of the original IAT, with participants classifying stimuli representing constructs of "death" and "life", and attributes them to "me" and "not me". A "D" score is calculated for each participant using reaction time. Positive D scores indicate a stronger association between death and self while negative scores represent a stronger association between life and self.
"Death/Life" Implicit Association Test. | One-month following treatment completion
  The d-IAT uses reaction time to measure automatic implicit associations with death and life stimuli. Procedures follow those of the original IAT, with participants classifying stimuli representing constructs of "death" and "life", and attributes them to "me" and "not me". A "D" score is calculated for each participant using reaction time. Positive D scores indicate a stronger association between death and self while negative scores represent a stronger association between life and self.

SECONDARY OUTCOMES:
Connection to Others | After treatment completion (week 4)
  The Interpersonal Needs Questionnaire (INQ-15) is a measure assessing beliefs about being a burden on others (i.e. perceived burdensomeness), and the extent to which an individual feels disconnected from others (i.e. thwarted belongingness). The scale is made up of a total of 15 items, six items assess for belongingness, and nine items measure burdensomeness. Responses are rated on a 7-point Likert-scale (1 = not at all true for me; 7 = very true for me), with higher scores reflecting higher levels of thwarted belongingness and perceived burdensomeness.
Religious and Spiritual Struggles | After treatment completion (week 4)
  The Religious and Spiritual Struggles Scale was developed as a self-report measure to assess supernatural, interpersonal, and intrapersonal struggles known as religious and spiritual struggles. The measure was developed to be relevant to an individual irrespective of their perceived level of religiosity and spirituality. The 26-item scale includes six subscales: Divine, Demonic, Interpersonal, Moral, Ultimate Meaning, and Doubt. Items are rated on a 5-point scale (1 = not at all/does not apply; 5 = a great deal). Higher scores indicate more religious and spiritual struggles.
Reasons for Living | After treatment completion (week 4)
  The Reasons For Living Scale is a 48-item self-report scale that assesses reasons for not dying by suicide. The scale includes six sub-scales, including survival and coping beliefs, responsibility to family, child-related concerns, fear of suicide, fear of social disapproval, and moral objections. Each item is rated on its importance on a 6-point scale (1 = not at all important; 6 = extremely important). Scale scores are the mean rating of each item set.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Gai, MS, Principal Investigator — Florida State University
Locations (1):
- Florida State Univeristy, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share IPD. Data sharing must be approved by funding sources.

REFERENCES:
- [Background] Franklin JC, Fox KR, Franklin CR, Kleiman EM, Ribeiro JD, Jaroszewski AC, Hooley JM, Nock MK. A brief mobile app reduces nonsuicidal and suicidal self-injury: Evidence from three randomized controlled trials. J Consult Clin Psychol. 2016 Jun;84(6):544-57. doi: 10.1037/ccp0000093. Epub 2016 Mar 28. PMID 27018530

DOCUMENTS (1):
  • Informed Consent Form (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT05541900/ICF_000.pdf